CLINICAL TRIAL: NCT07040865
Title: Randomized, Single-Blind, Monocentric, Non-Inferiority Trial of Gadopiclenol (Vueway®) Contrast Agent Performance vs. Gadobutrol (Gadovist®) in the Workup of Incidental Renal and Adrenal Findings
Brief Title: Randomized Comparison of Contrast Agents Gadopiclenol and Gadobutrol in the Workup of Incidental Renal and Adrenal Findings
Acronym: IRAF-WORKUP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BASEC 2025-00253; BASEC 2025-00253 (Other: Cantonal Ethics Committee Bern, Switzerland)
Record Dates: First submitted 2025-06-16; First posted 2025-06-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Suspect Renal and Adrenal Imaging Findings
MeSH Terms: interventions — gadobutrol; gadopiclenol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gadobutrol (control) (Active Comparator): 0.1 mmol/kg gadobutrol will be injected intravenously.
  Interventions: Drug: Gadobutrol (Gadovist/Gadavist)
- Gadopiclenol (Experimental): 0.05 mmol/kg gadopiclenol will be injected intravenously.
  Interventions: Drug: Gadopiclenol

INTERVENTIONS:
Drug: Gadobutrol (Gadovist/Gadavist) — Magnetic resonance acquisition without contrast agent followed the same acquisition 60 s and 15 min after gadobutrol contrast injection.
  Arms: Gadobutrol (control)
Drug: Gadopiclenol — Magnetic resonance acquisition without contrast agent followed the same acquisition 60 s and 15 min after gadopiclenol contrast injection.
  Arms: Gadopiclenol

SUMMARY:
The purpose of this study is to compare the effects of the contrast agent Gadopiclenol with those of the standard contrast agent Gadobutrol.

The main question of this study is :

Does gadopiclenol offer diagnostic properties that are equally effective as those of gadobutrol?

Participants will be:

* randomly assigned to one of two groups: the experimental group, which receives gadopiclenol, or the control group, which receives gadobutrol. Each participant is informed of their group allocation prior to the magnetic resonance imaging (MRI) scan.
* invited for a single MRI appointment lasting approximately 60 minutes

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age ≥18 years
* compatibility with magnetic resonance imaging
* planned workup of kidney incidental finding or adrenal incidental findings (or both)
* body mass index (BMI) < 31 kg/m2

Exclusion Criteria:

* patients with implants that might affect imaging parameters in the region under investigation, as judged by the principal investigator
* vulnerable individuals
* claustrophobic individuals
* individuals that are cognitively impaired or unable to understand the language
* pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Enhancement of the kidney and adrenal tissue | 60s and 15min after contrast injection during the one and only imaging session
  The primary endpoint is the enhancement of the kidney and adrenal tissue (difference of T1, longitudinal relaxation time, of the organ signal before and after contrast agent application) in both contrast agent groups 60s and 15min after contrast injection.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Christe, Prof. Dr. med., Principal Investigator — Bern University Hospital, Inselspital
Locations (1):
- Department of Diagnostic, Interventional and Pediatric Radiology Inselspital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol, including the case report form with the type of variables collected for each individual will be shared.
Supporting Information: Study Protocol
Time Frame: The Study Protocol will be made available at end of study. The availability will be open-ended.
Access Criteria: The IPD will be available to researchers, healthcare and patients through a yet to identify platform.